CLINICAL TRIAL: NCT06342232
Title: Study Protocol for a Randomized Controlled Trial on Neurofeedback Mindfulness and Its Efficacy on Migraine Management
Brief Title: The Efficacy of Neurofeedback Mindfulness in Migraine Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Marla Mickleborough, Dr. Marla Mickleborough, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEH1986; 423629 (Other Grant/Funding Number: Saskatchewan Health Research Foundation)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Migraine Headaches
Keywords: migraine; neurofeedback mindfulness; RCT
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback Mindfulness (Experimental): The participants received 8 weeks of intervention (10 min/day) including a neurofeedback mindfulness exercise via a portable EEG headband.
  Interventions: Behavioral: Neurofeedback mindfulness
- Simple Attention Task (Active Comparator): In the control group, the participants used the portable EEG headband for the same duration of intervention (8 weeks of practice, 10 min/day), but only listened to an audiobook without realtime access to their EEG recordings.
  Interventions: Behavioral: Simple attention controlled task

INTERVENTIONS:
Behavioral: Neurofeedback mindfulness — The participants used a portable EEG headband to complete 10 minutes of neurofeedback mindfulness practice for 8 weeks. While being seated comfortably, they could modify their brains rates based on the audio neurofeedback they received.
  Arms: Neurofeedback Mindfulness
Behavioral: Simple attention controlled task — The controlled group of this project also received an intervention which included an audiobook. While wearing the headband, the controlled participants muted their neurofeedback sounds and only focused on an audiobook while remaining relaxed. A summary of their brain states was given to them when completing their practice every day.
  Arms: Simple Attention Task

SUMMARY:
This longitudinal randomized controlled trial explored how long-term practice of neurofeedback mindfulness would be helpful for migraine management when compare dot a similar controlled intervention. All the participants went through assigned 10 minutes practices on a daily basis for 8 weeks. Behavioural reports and migraine characteristics were compared before and after the intervention.

DETAILED DESCRIPTION:
This study was announced on PAWS platform from September 2020 until December 2021 available for students, professors, employees and alumni at the University of Saskatchewan. Before the participant recruitment, 218 volunteers provided their consent and filled out the initial survey to be evaluated based on the study's criteria. The eligibility criteria included age, an official diagnosis of migraine from a clinician or meeting criteria for a migraine diagnosis based on ICHD-3 (2018), residing in Saskatoon area, having frequent headaches at least once a month, and access to smartphone and internet connection. A priori exclusion criteria for this study were comorbidity of Raynaud's syndrome or diabetes, frequent use of a preventative migraine treatment, and background experience with meditation.

After applying inclusion and exclusion criteria, participants were randomly selected for the NM or the control group. An invitation letter was sent to 112 volunteers (NM=53, control=59); out of which 11 individuals (NM=4, control=7) refused to participate due to different reasons (e.g., COVID-19, difficulty with device delivery, starting preventative medication or unstable migraine attacks) or never responded to the invitation or the follow up emails.

101 participants started the RCT (NM=49, control=52) but after attritions, 68 participants completed their total practice days. 4 participants in the control group were excluded from data analysis due to missing questionnaires and therefore insufficient data for repeated measures analysis. Three participants were also excluded due to inconsistency in their data or ethical considerations. As a result, we ended up having 61 participants (meditation=34, control=27) with complete intervention and available data for analysis. The mean average age was similar between the NM (age M= 34.11, SD= 9.89) and control groups (age M= 31.51, SD= 10.20). In the NM group, there were 28 females (82.4%) and 6 males (17.6%) and in the control group, we had 21 females (77.8%) and 6 males (22.2%). At the end of the study, the NM group had filled out 148 diaries, and the control group provided 100 diaries about their headaches.

Data collection occurred between September 2021 to December 2022 dependent on the joining date of each participant.

The initial questionnaire of this study included 45 open-ended and multiple-choice questions (26 min to complete) and was used to distinguish the inclusion and exclusion criteria. Having given the consent, the volunteers provided demographic information about their headache characteristics, family history of migraine headaches, and background experience with meditation.

After checking the availability criteria, the invited participants received a coded email information with a description of their practice, as well a copy of their consent form and contact information of a researcher in charge for device delivery. Before device delivery, the researchers checked COVID-19 self-screening measures.

A zoom meeting was scheduled (estimated for 30-60 minutes) after the participants would receive the device. In the initial meeting, the participants were introduced to focused listening and mind wandering states; they were suggested to block mind wandering during the sessions by attending to the audiobook carefully. Followed by the practice session, the participants would receive the same feedback of brain activities as shared by the NM group. The feedback included a timeline indicating their brain states (active, or relaxed) during the practice as well as reinforced consistent relaxed states. In this way, the control group task was identical to the NM group except that they listened to an audiobook instead of doing the NM intervention. For the whole duration of data collection (September 2021-December 2022), the sessions were monitored daily via MUSE Connect and were transcribed on an Excel file with information about numbers and reasons for missing days.

During the online session, participants received a brief introduction to the study goals and the participants' assigned task, and they were instructed on how to use the headband and the MUSE app to complete their given exercises both in the NM and control group. Participants were required to complete the pre-intervention questionnaire on the day of the initial meeting. After the initial meeting, they received daily reminders scheduled for 8:00 p.m. by a researcher. They were required to respond to the researcher by sending "1" for a complete session. Participants received a manual reply to keep them more engaged in the intervention. All the participants' practices were monitored daily via MUSE Connect. Information was collected about the duration of their practice, as well as the percentage of their relaxed or active states. In case of a pause in daily practices for more than three sessions, the researcher would send a follow up email asking for the reason of the pause in the intervention. In the event of having issues with the device, a EEG headband replacement was scheduled to be delivered to participants upon their availability. Additionally, the participants received weekly reminder text messages for headache diary questionnaires that were accessible via a SurveyMonkey link on their cellphones. Time to complete the diaries was estimated about 9 minutes, and the diaries included 24 multiple choices about subjects' recent headache experience.

On Week 8 of the study, the participants were given the post-intervention questionnaires to complete. In case of not completing the questionnaires, reminder emails were sent for 1 week.

Since this study was demanding and expected high amount of commitment for a long period of time, the participants' collaboration was appreciated by allowing them to keep their MUSE EEG headband at the end of the study after completion of the data. The participants who withdrew before completion were also allowed to keep their device.

Based on the rate of withdrawals and commitment to fill out the questionnaires, the attrition rate was 35.84% in the NM group and 54.23% in the control group; this made the total rate of attrition up to 39.60%. Since the rate of adherence to completing questionnaires and staying on task was different in the two groups, regardless of equal and balanced task requirements, this information is used as an indication of the interventions' feasibility and participants' adherence to the tasks.

We utilized five measurements, administered to participants before and after the study. On average, completing the five questionnaires was estimated to take about 13 minutes. These measurements collected information about migraine disability (MIDAS), headache severity (HIT-6), headache management self-efficacy (HMSE), anxiety (BAI), and depression (CES-D).

ELIGIBILITY:
Inclusion Criteria:

* age (over 18 years of age)
* a migraine diagnosis or having met the criteria for any type of migraine diagnosis based on ICHD-3 4. residing in Saskatoon or being able to receive the device from Saskatoon and the communities nearby
* having a smartphone and internet connection for accessing the MUSE app

Exclusion Criteria:

* Frequent background experience of meditation
* Comorbidity of Raynaud's syndrome or diabetes
* Current use of a preventative migraine treatment over 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Migraine Disability | 8 Weeks
  Based on MIDAS scale
Migraine Severity | 8 Weeks
  Based on Hit-6 Scale
Headache Management Self-efficacy | 8 Weeks
  Based on HMSE scale

SECONDARY OUTCOMES:
Anxiety | 8 Weeks
  Based on Beck Anxiety Index
Depression | 8 Weeks
  Based on CES-D scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No